CLINICAL TRIAL: NCT01273077
Title: Evaluation of Universal Rotavirus Vaccination Program
Status: Completed | Type: Observational
Sponsor: Dalhousie University (Other)
Collaborators: IWK Health Centre (Other); University of Prince Edward Island (Other); Horizon Health Care New Brunswick (Unknown); GlaxoSmithKline (Industry); Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Scott Halperin, Dr. Scott Halperin, Dalhousie University
Other Study IDs: GS1001; REB 4997 (Other Grant/Funding Number: GlaxoSmithKline); NCT01401686 (obsolete NCT alias)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Gastrointestinal Diseases
Keywords: Rotavirus; Rotarix
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Evaluation of Rotarix Program: All infants in Nova Scotia DHA 9 and PEI born after October1, 2010 until September 30, 2012 will be eligible for Rotarix immunization as part of the publicly funded immunization program. New Brunswick will serve as the non-intervention control location.
- Retrospective Surveillance: All laboratory- confirmed cases of rotavirus gastroenteritis and all cause diarrhea admitted to the trial hospitals from 2008-2010 will be entered in the database.
- Prospective Surveillance: Will begin on December 1, 2010. Data will be collected to identify hospitalizations for all cause diarrhea and rotavirus gastroenteritis at all 3 sites through the first two consecutive rotavirus seasons following vaccination.
- Safety Intussusception: Each trial hospital will identify cases of severe diarrhea and intussusception in Rotarix vaccine recipients through the first two consecutive rotavirus seasons following vaccination.
- ED Rotavirus Snap Shot Study: During rotavirus peak season, a prospective study of a sample of children under the age of 2 years presenting with diarrhea with or without vomiting to the ER of participating trial centers will be conducted in year one. In year 2 and 3 of the project:, systematic stool sampling will be carried out for cases of gastroenteritis in children < 5 years of age presenting to the ED departments.
- KAB Questionnaire for HCP and Parents: Data will be collected by a validated survey given to Parents, Healthcare providers and Program organizers throughout the 2 year program.

SUMMARY:
Two rotavirus vaccines have been authorized for use in Canada: RotaTeq®, Merck Frost Canada, Inc. and Rotarix®, Glaxo Smith Kline (GSK). In contrast to the United States, Australia and several other western countries, neither rotavirus vaccine is offered in a publicly funded program in Canada. A universal rotavirus immunization program offered to all children has the potential to prevent moderate to severe forms of the disease associated with rotavirus, with associated decreased disease burden and health care costs. This demonstration project seeks to evaluate the effect of the implementation of a universal infant immunization program with Rotarix employing two different program delivery models (public health delivery or physician office delivery) in comparison to a jurisdiction where routine immunization is not provided. Only evaluation of the program will be the subject of this study.

DETAILED DESCRIPTION:
Rotavirus immunization will be provided as part of the routine, publicly provided immunization program in PEI through Public Health Clinics and in Nova Scotia District Health Authority (DHA) 9 through physicians' offices. Saint John, New Brunswick will act as the control site where no publicly funded immunizations with Rotarix are provided. There are four components to the demonstration project which will take place at each of the three sites: retrospective surveillance, prospective surveillance, a prospective Emergency Department study, and an overall evaluation of the program and its acceptability. Actual provision of the vaccine through a universal immunization program will be undertaken by public health in PEI and in NS DHA 9. The objectives of the rotavirus surveillance (retrospective/prospective) and prospective ED study are:

1. To evaluate vaccine efficacy against rotavirus gastroenteritis of any severity in children under one - three year(s) of age following 2 oral doses of Rotarix.
2. To evaluate the burden of illness (hospitalization) associated with rotavirus infection in children less than 12 months - 3 years of age.
3. To monitor the incidence of severe side effects associated with uptake of Rotarix vaccine in program participants.
4. To provide data that is required to estimate costs associated with managing rotavirus in a hospital setting and at home.

The objectives for the universal rotavirus immunization program evaluation are:

1. To examine and compare the effectiveness of two program delivery systems (physician administered and public health administered) in providing the rotavirus vaccination to infants.
2. To evaluate the logistics of program implementation using the Rotarix vaccine in a cohort of infants.
3. To evaluate the acceptability of a universal rotavirus vaccination program by parents, physicians and nurses by measuring parent, nurse, and physician Knowledge Attitudes and Beliefs about rotavirus gastroenteritis.

ELIGIBILITY:
Rotarix immunization Program:

Inclusion criteria:

All infants in Nova Scotia DHA 9 and PEI born between October 1, 2010 and September 30, 2012. 6 weeks to 6 months of age at time of vaccination.

Exclusion:

* Infants who are hypersensitive to this drug or to any ingredient in the formulation or component of the container.
* Infants who experienced hypersensitivity after previous administration of rotavirus vaccines.
* Infants with uncorrected congenital malformation (such as Meckel's diverticulum) of the gastrointestinal tract that would predispose for intussusception.

Retrospective Surveillance (2008-2010)

Inclusion criteria:

* Confirmed rotavirus case in stool specimen taken within 14 days after the onset of gastrointestinal symptoms. Cases identified by autopsy must have had gastrointestinal symptoms before death.
* Rotavirus identified during 2008-2010
* Children less than 2 years of age
* Inpatient at site hospital
* Any patient who has a documented rotavirus hospital acquired infection
* Referred confirmed cases from another institution.

Exclusion Criteria:

* Non-laboratory confirmed diagnosis.
* Cases which do not have clinical data accessible by the nurse monitors

Prospective surveillance

Inclusion/Exclusion criteria:

Same as listed above for retrospective surveillance except the time period of surveillance will be December 1, 2010 - November 30, 2013.

Safety monitoring Intussusception Surveillance:

Inclusion criteria: Year 1 and 2

* Children less than 2 years of age presenting to the study site hospital (inpatients and outpatients)
* Radiologic or surgical diagnosis of intussusception and based on the Level 1 Brighton criteria:

  1.Invagination of the intestine (intussusception) demonstrated at surgery /2 demonstrated using air or liquid contrast enema 3.An intra-abdominal mass demonstrated using ultrasound or CT scan and was proven to be reduced by hydrostatic enema on a post-reduction imaging 4.Invagination of the intestine (intussusception) demonstrated at autopsy
* Presentation to hospital from December 1, 2010 - November 30. 2012

Exclusion criteria:

* Children 2 years of age or older
* Children with intussusception which is a direct complication of a surgical procedure.

  * Year 3 will include children less than 3 years of age

Emergency Department Rotavirus Snap Shot Study

Inclusion criteria: Year 1

* All children less than 2 years-old presenting with gastroenteritis who have a positive confirmed test for rotavirus, stool specimen taken within 14 days after the onset of symptoms.
* Telephone informed consent obtained from the parent or legal guardian.
* Parent or legal guardian can read and write English and can understand the informed consent documents and the study instructions and are mentally competent to give consent.

Exclusion Criteria:

* No stool sample
* Authorization not obtained

In year 2 and 3 of the project:, systematic stool sampling will be carried out for cases of gastroenteritis in children < 5 years of age presenting to the ED departments.

KAB Questionnaire for Health Care Providers and Parents

Inclusion criteria:

* Parents of healthy newborns eligible for the Rotarix vaccination program
* Parents who have a good understanding of English.
* Providers who were registered with the College of Registered Nurses of Nova Scotia, the Association of Registered Nurses of Prince Edward Island, the Nurses Association of New Brunswick, the Nova Scotia College of Family Physicians, the Prince Edward Island College of Family Physicians, or the New Brunswick College of Family Physicians for at least one year.
* Program managers responsible for immunization programs in PEI and NS DHA 9

Exclusion Criteria:

•Parents of newborns with a debilitating disease

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All infants in Nova Scotia DHA 9 and PEI born after October 1, 2010 until September 30, 2012 will be eligible for Rotarix immunization. Infants must be 6 weeks to 6 months of age at time of vaccination.
  All confirmed hospitalized Rotavirus cases from 2008-2010 and 2010-2013 will be entered in a database.
  All Intussusception cases after program start.
  Small sample size of outpatient confirmed rotavirus cases during rotavirus peak season 2011 and 2013 will be studied.
  Parents of infants eligible to receive Rotarix during the program will be invited to complete a KAB survey during the program as well as all healthcare providers eligible to administer Rotarix vaccine. Program organizers will be invited to take part in key informant interviews at the end of the program.
Sampling Method: Non-Probability Sample
Enrollment: 12705 (Actual)
Dates: Start 2010-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of Rotarix as detected through reduction of burden of illness due to rotavirus gastroenteritis | 2 years
  Our hypothesis for the first primary objective is that implementation of a universal rotavirus immunization program will result in a decreased burden of disease, as defined by number of hospitalizations in infants under one year of age, due to rotavirus. Evaluation of this objective will consist of the collection and comparison of retrospective and prospective surveillance data.

SECONDARY OUTCOMES:
To evaluate the implementation of a universal infant rotavirus immunization program with Rotarix | 2 years
  We do not have a hypothesis for the second primary objective as it is a descriptive analysis of program implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Donna MacDougall, PhD, RN, Principal Investigator — Canadian Center for Vaccinology
Locations (1):
- Canadian Center for Vaccinology, IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Zelman M, Sanford C, Neatby A, Halperin BA, MacDougall D, Rowswell C, Langley JM, Halperin SA; Maritime Universal Rotavirus Vaccination Program (MURVP). Implementation of a universal rotavirus vaccination program: comparison of two delivery systems. BMC Public Health. 2014 Sep 2;14:908. doi: 10.1186/1471-2458-14-908. PMID 25182067
- [Result] Sanford C, Langley JM, Halperin SA, Zelman M, Mvrvp. A universal infant rotavirus vaccine program in two delivery models: Effectiveness and adverse events following immunization. Hum Vaccin Immunother. 2015;11(4):870-4. doi: 10.1080/21645515.2015.1012028. PMID 25746110
- [Derived] MacDougall DM, Halperin BA, Langley JM, MacKinnon-Cameron D, Li L, Halperin SA; Maritime Universal Rotavirus Vaccination Program (MURVP). Knowledge, attitudes, beliefs, and behaviors of parents and healthcare providers before and after implementation of a universal rotavirus vaccination program. Vaccine. 2016 Jan 27;34(5):687-695. doi: 10.1016/j.vaccine.2015.09.089. Epub 2015 Oct 14. PMID 26458809
- See also: Canadian Center for Vaccinology — http://centerforvaccinology.ca
- See also: BMC Public Health.2014, 14:908 — http://www.biomedcentral.com/1471-2458/14/908